CLINICAL TRIAL: NCT07186673
Title: The Effectiveness of Using the Hall Technique in Restoring First Permanent Molars
Brief Title: Hall Technique vs Conventional Crown Restoration in Permanent Molars: Split-Mouth Trial in Children
Acronym: HTCC-SM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Hall T in Permanent Molars
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Permanent Molars; Dental Caries; Tooth Decay; Permanent First Molar Caries
Keywords: Hall Technique; Stainless Steel Crowns; Permanent First Molars; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Model Description:
  This is a randomized, controlled, split-mouth clinical trial in which each participant receives both interventions: the Hall Technique and the conventional crown preparation method. Each technique is applied to a different permanent first molar within the same child, allowing for direct within-subject comparison. Treatment allocation to the left or right molar is randomized. This design minimizes inter-individual variability and enhances the reliability of outcome comparisons.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Technique (Experimental): Permanent first molars are restored using the Hall Technique. No local anesthesia, caries removal, or tooth preparation is performed. Orthodontic separators are placed if needed, followed by stainless steel crown (SSC) cementation using glass ionomer cement.
  Interventions: Device: Stainless steel crown placement using Hall Technique
- Conventional Crown Preparation (Active Comparator): Permanent first molars are restored using the conventional method. Local anesthesia is administered, and the tooth is prepared with occlusal and proximal reduction before placement and cementation of a stainless steel crown using glass ionomer cement.
  Interventions: Device: Stainless steel crown placement using conventional method

INTERVENTIONS:
Device: Stainless steel crown placement using Hall Technique — Preformed stainless steel crowns are placed on permanent first molars without local anesthesia, caries removal, or tooth preparation. Orthodontic separators are used as needed, and crowns are cemented with glass ionomer cement
  Arms: Hall Technique
Device: Stainless steel crown placement using conventional method — Preformed stainless steel crowns are placed after administering local anesthesia and performing standard tooth preparation, including occlusal and proximal reduction. Crowns are cemented with glass ionomer cement.
  Arms: Conventional Crown Preparation

SUMMARY:
The aim of this study is to compare the clinical and radiographic success of stainless steel crowns placed using the Hall Technique versus the conventional method in the restoration of permanent first molars in children, and to evaluate their effects on occlusal relationships, crown adaptation, and patient satisfaction.

Study Outcomes The primary outcome of this study was to evaluate the clinical and radiographic success of stainless steel crowns placed on permanent first molars using the Hall Technique in comparison to the conventional crown placement method. The secondary outcomes included assessment of the marginal fit and adaptation of preformed crowns using both techniques, analysis of changes in occlusal relationships-specifically the vertical dimension of occlusion and overbite-and evaluation of patient satisfaction. Patient satisfaction was measured using a five-point Likert scale at multiple time points: immediately post-treatment, and at one, three, and six months.

DETAILED DESCRIPTION:
Detailed Description of the Study

This clinical study is designed to evaluate and compare the clinical and radiographic effectiveness of the Hall Technique and the conventional crown placement method for restoring permanent first molars in children using a split-mouth design. The study will be conducted at the Department of Pediatric Dentistry, Faculty of Dentistry, Tishreen University.

A total of 10 pediatric patients will be recruited according to specific inclusion and exclusion criteria. Each child will present with at least two eligible permanent first molars requiring full coronal restoration with stainless steel crowns. In the split-mouth design, each child will serve as their own control: one molar will be treated using the Hall Technique (HT), and the contralateral molar will be restored using the conventional method. The allocation of which technique will be applied to which side will be randomized for each patient to minimize bias.

Inclusion criteria will include:

* Permanent first molars with carious lesions affecting two or more surfaces or presenting Molar Incisor Hypomineralization (MIH).
* Absence of clinical signs or symptoms of irreversible pulpitis.
* Radiographic confirmation of an intact dentin layer and absence of internal or external root resorption or periapical pathology.

Exclusion criteria will include:

* Known allergy to nickel.
* Severely broken-down molars not suitable for SSC placement.
* Missing opposing teeth.
* Pulpal exposure during treatment.

In the HT group, stainless steel crowns will be placed without local anesthesia, without caries removal, and without any tooth preparation. Orthodontic separators will be placed if necessary during the first visit, and crown cementation will be performed using glass ionomer cement (GIC) during the follow-up visit.

In the conventional group, local anesthesia will be administered, and standard tooth preparation will be carried out (occlusal and proximal reduction), followed by fitting and cementation of the stainless steel crown using GIC.

Clinical and radiographic evaluations will be conducted at multiple time points: at baseline, 1 week, 1 month, 3 months, and 6 months post-treatment. These evaluations will aim to assess the success of the restoration based on crown integrity, presence of clinical symptoms, and radiographic signs of pulpal or periapical pathology.

Patient satisfaction will be measured using a five-point Likert scale, recorded immediately after treatment and again at 1 month, 3 months, and 6 months.

The primary outcome of the study will be the clinical and radiographic success of the restorations.

The secondary outcomes will include assessment of marginal fit and crown adaptation, changes in occlusal relationships (overbite), and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria (Clinical):

* No signs or symptoms of irreversible pulpitis
* Molars with carious lesions affecting two or more surfaces
* Permanent first molars with developmental defects

Inclusion Criteria (Radiographic):

* First molars with an intact dentin layer visible radiographically
* No signs of internal or external resorption
* No evidence of periradicular bone resorption

Exclusion Criteria:

* Patients with known nickel allergy
* Severely damaged molars not restorable with preformed crowns
* First molars without opposing teeth
* Pulp exposure during caries excavation

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Clinical and Radiographic Success | Baseline, 1 month, 3 months, and 6 months
  Clinical and Radiographic Success Definition: Absence of clinical symptoms (pain, swelling, mobility) and absence of radiographic signs of pathology (periapical radiolucency, internal/external resorption).

SECONDARY OUTCOMES:
- Marginal Fit and Adaptation - Changes in Occlusion ( Overbite) - Patient Satisfaction (Likert Scale) | Time Frame: Immediately post-treatment, 1 month, 3 months, and 6 months
  Secondary Outcome Measures
  Marginal Fit and Adaptation of Crown Definition: Clinical assessment of marginal adaptation (good, acceptable, poor).
  Time Frame: Post-treatment, 1 month, 3 months, and 6 months
  Changes in Occlusion (Overbite) Definition: Measurement of changes in vertical dimension of occlusion and overbite using clinical examination.
  Time Frame: Post-treatment, 1 month, 3 months, and 6 months
  Patient Satisfaction (Five-Point Likert Scale) Definition: Patient-reported satisfaction using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied). Higher scores indicate greater satisfaction.
  Time Frame: Immediately post-treatment, 1 month, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Study Chair — Tishreen University
Locations (1):
- Faculty of Dentistry, Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No
The decision regarding IPD sharing has not been finalized. Will follow institutional and regulatory guidelines.